CLINICAL TRIAL: NCT04267120
Title: A Single Arm, Multicenter, Phase 2 Trial to Evaluate the Efficacy of Lenvatinib (LEN) in Combination With Pembrolizumab (KEYtruda) in Subjects With Locally Advanced or Metastatic Non-clear Cell Renal Cell Carcinoma (The LENKYN Trial)
Brief Title: Lenvatinib (LEN) in Combination With Pembrolizumab (KEYtruda) in Subjects With Locally Advanced or Metastatic Non-clear Cell Renal Cell Carcinoma (The LENKYN Trial)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment with low accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202003148
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lenvatinib + Pembrolizumab (Experimental): * Lenvatinib 20 mg/day will be administered orally on a daily basis and pembrolizumab 200 mg will be infused once every 3 weeks.
  * Subjects may be treated with pembrolizumab for a maximum of 35 cycles or approximately 2 years, but treatment with lenvatinib can continue beyond 2 years if the subject does not meet other treatment discontinuation criteria.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab; Procedure: Research blood collection

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be provided by Merck.
  Other Names: Lenvima; Lenvanix
Drug: Pembrolizumab — Merck will provide pembrolizumab
  Other Names: Keytruda; MK-3475
Procedure: Research blood collection — -Within 2 weeks prior to first dose of study drug, cycle 4 day 1, and at the off-treatment assessment

SUMMARY:
This is a single-arm, multicenter, phase 2 study of lenvatinib in combination with pembrolizumab (lenvatinib 20 mg/day + pembrolizumab 200mg q3weeks) in subjects with unresectable advanced or metastatic non-clear cell renal carcinoma who have not received any chemotherapy for advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic histologically confirmed nccRCC (2, 7). Must have one of the following subtypes of nccRCC:

  * papillary RCC
  * chromophobe RCC
  * TFE-3/B translocation RCC
  * SDHB-loss RCC
  * TSC1-loss RCC
  * sarcomatoid RCC without clear cell component
  * unclassified RCC
* Has not received any prior lines of systemic therapy except adjuvant or neoadjuvant treatments.
* Radiologically measurable disease meeting the following criteria:

  * At least 1 lesion of ≥ 10 mm in the longest diameter for a non-lymph node or ≥ 15 mm in the short axis diameter for a lymph node which is serially measurable according to iRECIST (Section 12) using computerized tomography (CT) or magnetic resonance imaging (MRI).
  * Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of subsequent progressive disease (substantial size increase of ≥20%) to be deemed a target lesion. Patients who received EBRT must be at least 2 weeks out from last RT treatment.
* At least 18 years of age.
* Karnofsky performance status ≥ 70%
* Blood pressure (BP) ≤ 150/90 mmHg at screening with or without antihypertensive medications and no change in antihypertensive medications within 1 week prior to Cycle 1 Day 1.
* Adequate renal function defined as creatinine <1.5 x ULN or calculated creatinine clearance ≥40 mL/min per the Cockcroft and Gault formula with creatinine levels >1.5 x ULN.
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) ≥1500/mm3 (≥1.5 x 103/L)
  * Platelets ≥100,000/mm3 (≥100 x 109/L)
  * Hemoglobin ≥9.0 g/dL
* Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) ≤1.5
* Adequate liver function as evidenced by:

  * bilirubin ≤1.5 times the upper limit of normal (ULN)
  * alkaline phosphatase (ALP) ≤3×ULN (in the case of liver metastases ≤5×ULN)
  * alanine aminotransferase (ALT) ≤3×ULN (in the case of liver metastases ≤5×ULN)
  * aspartate aminotransferase (AST) ≤3×ULN (in the case of liver metastases ≤5×ULN).

In case ALP is >3×ULN (in the absence of liver metastases) or >5×ULN (in the presence of liver metastases) AND the subject also is known to have bone metastases, the liver specific ALP isoenzyme must be separated from the total and used to assess the liver function instead of the total ALP.

* Subjects with known brain metastases will be eligible if they have completed the primary brain therapy (such as whole brain radiotherapy, stereotactic radiosurgery, or complete surgical resection) and if they have remained clinically stable, asymptomatic, and off steroids for at least 2 months before starting study treatment.
* All females of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta-human chorionic gonadotropin [β-hCG]) at the screening visit. Females of childbearing potential* must agree to use a highly effective method of contraception for the entire study period and for 120 days after study discontinuation
* Male subjects who are partners of women of childbearing potential must follow one of the methods of contraception described in Section 6.5 beginning at least 1 menstrual cycle prior to starting study drugs, throughout the entire study period, and for 120 days after the last dose of study drug, unless the male subjects are totally sexually abstinent or have undergone a successful vasectomy with confirmed azoospermia or unless the female partners have been sterilized surgically or are otherwise proven sterile.
* Archival tumor tissue from within 3 months (preferred) or up to 6 months (acceptable) must be available prior to the first dose of study drug for biomarker analysis. If no biopsy has been performed in the prior 6 months, a standard of care biopsy is requested if safe and feasible. In the case tissue cannot be provided, patients can be enrolled upon consultation and agreement by the trial PI.

Note: In case of submitting unstained cut slides, freshly cut slides should be submitted to the testing laboratory within 14 days from when the slides are cut.

-Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Predominant clear cell renal cell carcinoma (RCC)
* Uncontrolled or untreated brain metastasis
* Major surgery performed within 4 weeks prior to the first dose of study drugs or scheduled for major surgery during the study. Subjects must have recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy.
* Subjects having >1+ proteinuria on urinalysis will undergo 24-h urine collection for quantitative assessment of proteinuria. Subjects with urine protein ≥1 g/24-hour will be ineligible.
* Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
* New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months.
* Prolongation of QTc interval to >480 msec.
* Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
* Active infection (any infection requiring systemic treatment).
* Subject is known to be positive for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
* Serious nonhealing wound, ulcer, or bone fracture.
* Known intolerance to either of the study drugs (or any of the excipients).
* History of organ allograft (subject has had an allogenic tissue/solid organ transplant) or allogeneic stem cell transplant (subject has received blood-forming stem cells from a donor).
* Biologic response modifiers (e.g., granulocyte colony-stimulating factor) within 4 weeks before study entry. Chronic erythropoietin therapy is permitted provided that no dose adjustments were made within 2 months before first dose of study treatment.
* Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment. If the required urine pregnancy test is positive (or cannot be confirmed as negative) within 72 hours prior to start of treatment, a serum pregnancy test will be required.
* Excluding the primary tumor leading to enrollment in this study, any other active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the bladder or cervix) within the past 36 months.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of up to 10 mg/day of prednisone or equivalent is approved and does not exclude the patient from the trial.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, > 10 mg of prednisone per day, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. The use of up to 10 mg/day of prednisone or equivalent is approved and does not exclude the patient from the trial.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required maintenance steroids (>10 mg of prednisone) or current pneumonitis/interstitial lung disease.
* Has received a live-virus vaccination or live-attenuated vaccine within 30 days of planned treatment start. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Picus, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Stanford Cancer Center, Palo Alto, California
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months after publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenvatinib + Pembrolizumab
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 57 [37 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: * ORR is defined as the proportion of subjects who have a best overall response of complete response (CR) or partial response (PR)
  * CR: Disappearance of target and non-target lesions and normalization of tumor markers.
  * PR: At least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the baseline sum of diameters. Non target lesions must be non-progressive disease.
Time Frame: Through completion of treatment (median length 287 days, full range 92-728 days)
Population: One patient was not evaluable as they did not have a disease assessment outside of the baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 10
Participants | 4

2. Secondary Outcome: Safety and Tolerability of Regimen as Measured by Related Adverse Events Experienced by Participant
Description: -Will be graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Time Frame: From start of treatment through 120 days after last day of study treatment (median length of follow-up 397 days, full range 92-848 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
Participants
  Abdominal pain | 2
  Adrenal insufficiency | 1
  Alanine aminotransferase increased | 1
  Alopecia | 1
  Anemia | 3
  Anorexia | 5
  Aspartate aminotransferase increased | 3
  Cholesterol high | 1
  Cognitive disturbance | 1
  Constipation | 1
  Creatinine increased | 1
  Depression | 1
  Diarrhea | 6
  Dizziness | 1
  Dry skin | 2
  Dysgeusia | 1
  Dysphagia | 1
  Enterocolitis infectious | 1
  Eosinophilia | 1
  Erythematous rash | 1
  Fatigue | 6
  Fecal incontinence | 1
  Generalized edema | 1
  Headache | 3
  Hemorrhoids | 1
  Hernia surgery | 1
  Hoarseness | 2
  Hypertension | 6
  Hyperthyroidism | 1
  Ileus | 1
  Incisional hernia | 1
  Insomnia | 1
  Intra-abdominal hemorrhage | 1
  Itchy scalp | 1
  Jejunal fistula | 1
  Mucositis oral | 2
  Myalgia | 1
  Nail discoloration | 1
  Nausea | 6
  Neutrophil count decreased | 2
  Non-cardiac chest pain | 1
  Pain - bottoms of feet | 1
  Palmar-plantar erythrodysesthesia syndrome | 5
  Papulopustular rash | 1
  Peripheral sensory neuropathy | 1
  Platelet count decreased | 1
  Proteinuria | 4
  Pruritus | 2
  Pruritic Rash | 1
  Rash | 1
  Rash acneiform | 1
  Rash maculo-papular | 2
  Restless Leg Syndrome | 1
  Scalp sores | 1
  Sensitive Hands | 1
  Sensitive skin/sores on face | 1
  Skin Soreness | 1
  Sore throat | 2
  Stomach pain | 1
  Thyroid stimulating hormone increased | 8
  Vision decreased | 1
  Vitiligo | 1
  Voice alteration | 1
  Vomiting | 3
  Warm hands and feet | 1
  White blood cell decreased | 1
  Weight loss | 2

3. Secondary Outcome: Cumulative Probability of Progression-free Survival (PFS)
Description: * PFS is defined as the time from date of first dose of study drug to date of first documentation of disease progression or death, whichever occurs first.
  * Progressive disease: At least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) AND an absolute increase of ≥5 mm. Appearance of new lesions will also constitute PD (including lesions in previously unassessed areas).
  * Cumulative probability is on a scale of 0-1.
Time Frame: At 3 months
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
probability | 1.0000 [1.0000 to 1.0000]

4. Secondary Outcome: Cumulative Probability of Progression-free Survival (PFS)
Description: * PFS is defined as the time from date of first dose of study drug t date of first documentation of disease progression or death, whichever occurs first.
  * Progressive disease: At least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) AND an absolute increase of ≥5 mm. Appearance of new lesions will also constitute PD (including lesions in previously unassessed areas).
  * Cumulative probability is on a scale of 0-1.
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
probability | 0.9091 [0.5081 to 0.9867]

5. Secondary Outcome: Cumulative Probability of Progression-free Survival (PFS)
Description: as for outcome 4
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
probability | 0.7273 [0.3708 to 0.9028]

6. Secondary Outcome: Median Progression-free Survival (PFS)
Description: * PFS is defined as the time from date of first dose of study drug to date of first documentation of disease progression or death, whichever occurs first.
  * Progressive disease: At least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) AND an absolute increase of ≥5 mm. Appearance of new lesions will also constitute PD (including lesions in previously unassessed areas).
Time Frame: Through completion of follow-up (median length 602 days, full range 92-1244 days)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
months | 19.78 [8.71 to 22.47]

7. Secondary Outcome: Median Overall Survival (OS)
Description: -OS is defined as the time from the date of first dose of study drug until date of death from any cause.
Time Frame: Through completion of follow-up (median length 602 days, full range 92-1244 days)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
months | 19.78 [11.43 to 36.53]

8. Secondary Outcome: Cumulative Probability of Overall Survival (OS)
Description: * OS is defined as the time from the date of first dose of study drug until date of death from any cause.
  * Cumulative probability is on a scale of 0-1.
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
probability | 0.9091 [0.5081 to 0.9867]

9. Secondary Outcome: Cumulative Probability of Overall Survival (OS)
Description: as for outcome 8
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
probability | 0.8182 [0.4474 to 0.9512]

10. Secondary Outcome: Cumulative Probability of Overall Survival (OS)
Description: as for outcome 8
Time Frame: At 18 months
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 11
probability | 0.6364 [0.2969 to 0.8452]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 120 days after last day of study treatment (median length of follow-up 397 days, full range 92-848 days). All-cause mortality was collected from start of treatment through completion of follow-up (median length 602 days, full range 92-1244 days).
Arm/Group | Lenvatinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 8/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib + Pembrolizumab (N=11)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac troponin I increased (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Jejunal fistula (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
New prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib + Pembrolizumab (N=11)
Anemia (Blood and lymphatic system disorders) | 6
Eosinophilia (Blood and lymphatic system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Adrenal insuffciency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Vision decreased (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Dental pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Pain - bottom of feet (General disorders) | 1
Chills (General disorders) | 2
Edema limbs (General disorders) | 2
Facial abrasions (General disorders) | 1
Fatigue (General disorders) | 9
Generalized edema (General disorders) | 1
Malaise (General disorders) | 1
Sweating (General disorders) | 1
COVID-19 infection (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 5
Blood bicarbonate increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 4
INR increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Thyroid stimulating hormone increased (Investigations) | 8
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Hip pain (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 2
Restless leg syndrome (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 5
Amenorrhea (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythematous rash (Skin and subcutaneous tissue disorders) | 1
Face sores (Skin and subcutaneous tissue disorders) | 1
Itchy scalp (Skin and subcutaneous tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Pruritic rash (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Scalp sores (Skin and subcutaneous tissue disorders) | 1
Sensitive hands (Skin and subcutaneous tissue disorders) | 1
Sensitive skin (Skin and subcutaneous tissue disorders) | 1
Skin soreness (Skin and subcutaneous tissue disorders) | 1
Sores above pubis area (Skin and subcutaneous tissue disorders) | 1
Warm hands and feet (Skin and subcutaneous tissue disorders) | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 1
Hernia surgery (Surgical and medical procedures) | 1
Incisional hernia (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT04267120/Prot_SAP_000.pdf